CLINICAL TRIAL: NCT06684873
Title: A Multicenter, Single-arm, Open-label Study Evaluating the Safety and Efficacy of AK112 Combined With Chemotherapy as First-line Treatment for Non-squamous NSCLC Patients With BRAIN Metastases and Negative Driver Genes (IVO BRAIN)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li-kun Chen, senior doctor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK112-IIT-C-M-0005
Record Dates: First submitted 2024-11-10; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: NSCLC; Brain Metastasases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK112 combined with chemotherapy (Experimental): AK112 combined with chemotherapy
  Interventions: Drug: AK112 Injection

INTERVENTIONS:
Drug: AK112 Injection — AK112 injection plus chemotherapy was administered to all eligible patients

SUMMARY:
A multicenter, single-arm, open-label study evaluating the safety and efficacy of AK112 combined with chemotherapy as first-line treatment for non-squamous NSCLC patients with BRAIN metastases and negative driver genes

DETAILED DESCRIPTION:
This is a multicenter, single-arm, open-label study. We planned to enroll 55 patients with histopathologically or cytologically confirmed stage IV nsqNSCLC with brain metastases and negative driver gene reports within three months. The aim of this study is to evaluate the safety, tolerability and efficacy of ivoricizumab combined with chemotherapy as the first-line treatment for patients with brain metastases from NSQ non-small cell lung cancer (NSCLC) without driver genes.

Eligible subjects were selected and entered the study in sequence. The trial was divided into combination chemotherapy period (C1-C4/C6) and maintenance treatment period (C5/C7-C32). During the combined chemotherapy period, all subjects were treated with everciximab injection and chemotherapy drugs after entering the study, and during the maintenance treatment period, they were treated with everciximab injection and pemetrexed. Every 3 weeks (Q3W) was a treatment cycle. The efficacy was evaluated every 2 cycles in the combined chemotherapy period and every 3 cycles in the maintenance treatment period. All the participants received treatment until they withdrew consent, had disease progression, had unacceptable toxicity, had to discontinue the drug as judged by the investigator, were lost to follow-up, died, or had received ivorximab for 2 years, whichever occurred first. After the end of treatment, the patients were followed up until death.

If there are abnormal items, for the safety of subjects, researchers can judge whether to add unplanned follow-up according to the actual situation.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily participated in the clinical study and had not received any systemic anti-tumor treatment (including any chemotherapy, targeted therapy, immunotherapy, etc.)
2. Male or female subjects aged 18-75 years (including the cutoff) at the time of signing the ICF
3. patients with histopathologically or cytologically confirmed stage IV non-squamous non-small cell lung cancer (nsqNSCLC) with brain metastases
4. Patients were required to provide a genetic testing report that showed negative driver genes, i.e., no EFGR sensitive gene mutation, no ALK or ROS1 gene fusion, no BRAF V600E sensitive gene mutation, and no RET gene fusion

5. If not, qualified tumor tissue or blood should be provided for genetic testing. 5) MRI confirmed brain parenchymal metastasis, with ≥3 brain lesions

6: Or patients with 1-2 brain lesions who are not suitable for local treatment or refuse local treatment. At least one measurable brain lesion had to be at least 5mm in diameter. 6) For asymptomatic brain metastases or those with controlled intracranial hypertension after treatment with dehydration, medication could be continued at enrollment or during the study to maintain symptom stability

7) At least one measurable target lesion as assessed by investigator according to RECIST v1.1 within 4 weeks before the first dose

8) ECOG PS score of 0-1

9) predicted survival time ≥12 weeks

10) good vital organ function

11) Female subjects must have a negative serum pregnancy test within 3 days before treatment, agree to use effective contraception during and after treatment for 6 months, and refrain from breastfeeding during treatment

12: Male patients provided consent to use contraception during treatment.

Exclusion Criteria:1) known history of severe allergy to any monoclonal antibody (NCI-CTCAE 5.0 > 3) Or known hypersensitivity to carboplatin/pemetrexed components

2: any active infection requiring systemic anti-infective therapy within 14 days before the first dose

3) myocardial infarction with uncontrolled arrhythmia (including QTc interval ≥450 ms in men and ≥470 ms in women) within 6 months before the first dose (QTc interval was calculated with Fridericia's formula)

4: Or grade III-IV cardiac dysfunction according to the New York Heart Association (NYHA) standard or left ventricular ejection fraction <50% by echocardiography

5) subjects with ≥ grade 2 CTCAE peripheral neuropathy

6) subjects had uncontrolled or symptomatic hypercalcemia (>1.5 mmol/L ionized calcium or calcium >12 mg/dL or corrected serum calcium >ULN)

7) subjects with previous or screening history of interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, or severely impaired pulmonary function, which may interfere with the detection and treatment of suspected drug-related pulmonary toxicity according to the investigator's judgment

8) untreated active hepatitis B subjects (HBsag-positive and HBV-DNA > 1000 copies /mL (200 IU/mL) or higher than the lower limit of detection, whichever is higher) and, for those with hepatitis B, required to receive anti-HBV treatment for the duration of the study treatment

9: Active hepatitis C subjects (positive for HCV antibodies and HCV-RNA levels above the lower limit of detection)

10: Or patients with known active syphilis infection (excluding patients with positive heterologous antibody test, negative non-heterologous antibody test and inactive infection confirmed by clinical judgment)

11 Or a known history of human immunodeficiency virus (HIV) positivity or screening positive for HIV

12) the subject has a known active or suspected autoimmune disease. Subjects who were in a stable state and did not require systemic immunosuppressive therapy were allowed to enroll.

13) patients with other active malignant tumors within 5 years or at the same time. Localized tumors that had been cured for more than 5 years, such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, prostate cancer in situ, cervical cancer in situ, and breast cancer in situ, were eligible for inclusion.

14) Recipients of a live or attenuated vaccine within 28 days before the first dose, or having a plan to receive such vaccine during the study period. However, inactivated virus vaccines for seasonal influenza are permitted

15) radical radiotherapy or whole brain radiotherapy (WBRT) to the skull within 3 months before the first dose

16) subjects with spinal cord compression that could not be cured by surgery and/or radiotherapy

17) patients with deep vein thrombosis, current anticoagulant or platelet therapy, or previous use of antiangiogenic drugs for deep vein thrombosis or severe bleeding

18) poorly controlled (poorly controlled defined as BP ≥160/100 MMHG despite optimal hypertension treatment)

19) had undergone major surgery within 28 days before the first dose (major surgery was defined for this study as a procedure requiring at least 3 weeks of recovery before being able to undergo study treatment)

20) who are participating in another clinical study, or who have participated in any other clinical trial (including drugs, devices, etc.) and received intervention within 3 months before screening or within 5 half-lives (whichever is longer)

21) candidates for or prior recipients of organ or bone marrow transplantation

22) subjects had a known history of psychotropic drug abuse or drug use

23) subjects with any factors considered by the investigator to be ineligible for the trial.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-11-02 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
iPFS | iPFS was defined as the time from the date of initiation of firstline setting to the date of intracranial progression or death and was censored at the date of the last tumor assessment (when carried out)
  iPFS was defined as the time from the date of initiation of firstline setting to the date of intracranial progression or death and was censored at the date of the last tumor assessment (when carried out)

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hou X, Li M, Wu G, Feng W, Su J, Jiang H, Jiang G, Chen J, Zhang B, You Z, Liu Q, Chen L. Gefitinib Plus Chemotherapy vs Gefitinib Alone in Untreated EGFR-Mutant Non-Small Cell Lung Cancer in Patients With Brain Metastases: The GAP BRAIN Open-Label, Randomized, Multicenter, Phase 3 Study. JAMA Netw Open. 2023 Feb 1;6(2):e2255050. doi: 10.1001/jamanetworkopen.2022.55050. PMID 36753281